CLINICAL TRIAL: NCT03291730
Title: A Nurse Led Project to Introduce Hand Lettering as a Form of Creative Art Expression to Patients in an Ambulatory Oncology Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Cindy L. Cao, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 17-377
Record Dates: First submitted 2017-09-20; First posted 2017-09-25 (Actual); Last update posted 2018-12-03 (Actual); Status verified 2018-11

CONDITIONS: Anxiety
Keywords: Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Respiration; Art Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hand Lettering (Experimental): * The participant will engage in art-therapy by tracing and coloring a detailed letter or word
  * Participants will also be guided through a relaxation breathing and journaling exercise that can be incorporated into the art activity.
  Interventions: Behavioral: Breathing and journaling exercise; Other: Art-therapy

INTERVENTIONS:
Behavioral: Breathing and journaling exercise — May help reduce anxiety of receiving chemotherapy
Other: Art-therapy — May help reduce anxiety of receiving chemotherapy

SUMMARY:
The investigators are conducting a project to provide a new type of resource called "hand lettering" to patients receiving chemotherapy. This is a type of art therapy. The goal of this project is to understand if it is feasible to use art-therapy and to describe anxiety before and after completing hand-lettering.

DETAILED DESCRIPTION:
This study is being done to understand if it is feasible to use a form of art-therapy called hand-lettering at Dana-Farber Cancer Institute. We would also like to explore the anxiety a person has before and after using hand-lettering.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>age 18) with a cancer diagnosis receiving oral or IV chemotherapy at Dana-Farber on Yawkey 10.
* Able to read and speak English
* Has a minimum appointment time of 60 minutes

Exclusion Criteria:

-Individuals with visual impairment or blindness will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-01-09 (Actual); Primary Completion 2018-06-05 (Actual); Study Completion 2018-06-05 (Actual)

PRIMARY OUTCOMES:
Evaluate the feasibility of implementing nurse-led hand-lettering in an ambulatory infusion setting | 2 years
  Feasibility will be defined through enrollment and completion rates.

SECONDARY OUTCOMES:
Describe patient self-reported anxiety before and after utilizing hand-lettering | 2 years
  Anxiety measured through the State Trait Anxiety Index.

CONTACTS AND LOCATIONS:
Overall Officials: Cindy L Cao, RN, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No